CLINICAL TRIAL: NCT06569628
Title: Validation Study of the Implementation of Narrative Care Methodology, Life Stories and Biographies in Long-Term Care Centres for Old-Adults
Brief Title: Validation of a Life Stories Methodologies in Long-Term Care Centres
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Envita Digital Solutions S.L. (Other)
Collaborators: Agencia Gallega de Innovación (GAIN) (Unknown); Faculty of Psychology, University of Santiago de Compostela, Santiago de Compostela, Galicia-Spain (Unknown); DomusVi, long-term care centres for old adults (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03_IN606D_2023_ 2529780
Record Dates: First submitted 2024-07-31; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Long-term Care Centres for Old Adults Users; Relatives of Long-term Care Centres for Old Adults Users; Long-term Care Centres for Old Adults Professionals
Keywords: Life Review; Life Story; Narrative Care; Digitalization; Envita Stories; Person-centred Care; Long-term Care Centres; Long-term Care

STUDY DESIGN:
Intervention Model Description: Long-term Care Centres for old adults users will be divided into three groups: 1)Intervention group: participates directly in the incorporation of the proposed methodology; 2)Contact group: participates indirectly (implementation of the methodology in the centres in which they reside but not in them directly); 3)Non-contact control group: resides in a centre in which the methodology is not being implemented. This process will also involve the reference professionals involved in the implementation of the methodology and those family members who voluntarily become involved in the care of the participants based on this methodology.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group in Long-term Care Centres for old adults (Experimental): This group participates directly in the incorporation of narrative care through the implementation of life stories and biographies (Envita Stories Methodology) in the long-term care centres for old adults in where they reside, through the specific workshops and by preparing their own life stories
  Interventions: Combination Product: Envita Stories Methodology in Long-term care Centres for old adults
- Contact group in long-term care Centres for old adults (Active Comparator): This group participates indirectly, through the implementation of the Envita Stories Methodology in the long-term care centres for old adults in which they reside but not in them directly
  Interventions: Behavioral: Contact Methodology in Long-term Care Centres for old adults
- Control group in Long-term care centres for old adults (No Intervention): This Group resides in a long-term care centres for old adults in which the methodology is not being implemented, although it will be implemented throughout the project process

INTERVENTIONS:
Combination Product: Envita Stories Methodology in Long-term care Centres for old adults — Collaborative intervention program in long-term care Centres for old adults between professionals, old adults, families and volunteers that aims to foster person-centered care and promote meaningful relationships through the digitization of life stories and life project methodologies in a timeline.
  Arms: Intervention group in Long-term Care Centres for old adults
Behavioral: Contact Methodology in Long-term Care Centres for old adults — Professionals know and use Envita Stories Methodology but do not apply it directly with these people.
  Arms: Contact group in long-term care Centres for old adults

SUMMARY:
The objective of the research is to validate a methodology for implementing narrative care, through the incorporation of people's biographies and life stories, in interventions in long-term care centres for older adults.

From a positivist perspective of gerontological intervention, priority will be given to the validation of quantitative methodologies with empirical support. The study will involve 378 users residing in Galician long-term care centres for older adults. At the theoretical level, there is a broad consensus among professionals and experts on the need to develop new methodologies that allow the personalization of long-term care care and facilitate the development and promotion of the life projects of the older persons through the provision of the support that a particular person needs. In addition, there is a large body of practical interventions that attempt to apply these postulates. However, there is a clear lack of research methodologies that provide robust scientific results and data to support and evaluate these new developments.

DETAILED DESCRIPTION:
A. Background

Narrative care and the methodology of incorporating biographies and life stories emerged in the context of long-term care centres for old-adults in response to the need to promote the deinstitutionalization of care and to advance in the transformation of the long-term care model towards a humanistic approach, and from the ethical and intervention proposal of person-centered care.

Putting this care approach into practice can be complex. In general, the traditional care model and seeing gerontological centers as "institutions" does not favor the implementation of person-centered care methodologies. Society, in general, and professionals in particular are faced with the challenge of promoting the search for solutions to care from a more human point of view in which the so-called "narrative care" takes center stage.

In this context, the need emerges to provide care professionals with new digital tools that facilitate the implementation of valuable methodologies such as life stories, the life project, the professional of reference and the support group, and develop proposals focused on favoring spaces for the creation and strengthening of bonds and meaningful relationships that promote the participation and social inclusion of the person in his/her environment and community, as a protective factor against unwanted loneliness in people in need of long-term care.

Furthermore, at the theoretical level, there is a broad consensus among professionals and experts on the need to develop new methodologies that allow the personalization of long-term care and facilitate the development and promotion of the life projects of the older persons through the provision of the support that a particular person needs. In addition, there is a large body of practical interventions that attempt to apply these postulates. However, there is a clear lack of research methodologies that provide robust scientific results and data to support and evaluate these new developments.

B. Problem or need to which it is intended to provide an answer.

This project jointly addresses the binomial long-term care-unwanted loneliness in long-term care centres for old-adults, betting on digitization as a key element in the search for solutions. The purpose is to advance the line of research in three main areas:

1. Narrative care and person-centered care

   Person-centered care (PCC) proposes a paradigm shift in long-term care, placing people in need of care/support and their life projects at the center of organizations, at the backbone of their processes.

   The life stories and the life project are advanced methodologies typical of person-centered care approaches that facilitate old-adults, in this case, are the axis around which the interventions and the day-to-day communications of the centers revolve.

   The professionals who care for and/or accompany people have to understand life stories method as the essence of person-centered care and humanization. The experts argue that it is an inexcusable component of genuine person-centered care, a component that acquires meaning not only by virtue of its effectiveness and the practical benefits it implies, but also as an ethical imperative of care. It is a valuable tool that allows us to know and recognize the person, to respect and understand him or her better.
2. Unwanted loneliness

   According to data from the survey on loneliness in older people conducted by La Caixa Foundation in 2018 in Spain, there is a higher prevalence of loneliness in institutionalized old adults than in the general population, with this prevalence being much higher.

   Another noteworthy fact is the high prevalence of institutionalized old adults who indicate that their life is not satisfactory and/or they do not feel that they have a meaningful life.

   In turn, most old adults feel unwanted loneliness throughout their lives, regardless of their living situation.

   The experts point out that the main interventions to alleviate loneliness are aimed at: 1) direct interventions with the person, fostering social connections and helping to maintain those that already exist; 2) interventions in the environment, focused on developing appropriate structural facilitators in a close environment to help reduce loneliness and prevent it in people at risk of experiencing it.
3. Digitalization

This project will offer an essential digital solution that guides, facilitates and supports the implementation of life stories and life project methodologies, through which it intervenes in 3 key concepts: 1) Care (personalized attention); 2) Involvement (meaningful activities, promotion of the life project); 3) Unwanted loneliness (creating spaces for valuable interactions and meaningful relationships), from the approach of good practice in the incorporation of technology in the field of care (Liedo and Ausín, 2022).

C. Objectives

The general objective is to empirically support the implementation methodology of narrative care by incorporating biographies and life stories in the context of long-term care with old adults, professionals and families, validating the effects of the program in centres.

The proposal would have two main specific objectives:

1. To review the empirical evidence on digital applications in PCC concepts.

   1.1. Care (personalization, personalized care) (Incorporation of biography into care).

   1.2. Involvement (Meaningful activities) (Promoting life project)

   1.3. Unwanted loneliness (relationships, bonds, community) (Create spaces for valuable interactions and meaningful relationships).
2. To validate the effects of the application of narrative care through the incorporation of life stories and biographies, in long-term care centres for old adults, by means of a randomized clinical trial.

2.1. To validate the cognitive effects of the application in long-term care centres for old adults.

2.2. To validate the functional impact of the application in long-term care centres for old adults, through the facilitation of participation in daily life and in their community and the promotion of new illusions, goals or dreams to be fulfilled.

2.3. To validate the effects at the affective level of the application in long-term care centres for old adults, through the promotion of emotional connection and the promotion of meaningful relationships.

2.4. To validate the effects on social support of the application in long-term care centres for old adults, through the activation of meaningful relationships, the strengthening of bonds and relationships of trust, encouraging family participation in care and improving communication patterns.

2.5. To assess the perception of professionals on the use of the resources deployed through the intervention methodology.

ELIGIBILITY:
Inclusion criteria: Old adults living in a long-term care centre in Galicia (Spain).

Exclusion criteria: N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive status | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  Montreal cognitive assessment (MoCA). The Montreal Cognitive Assessment (MoCA) is designed to assess mild cognitive dysfunction. This instrument examines the following skills: attention, concentration, executive functions (including the capacity for abstraction), memory, language, visuoconstructive abilities, calculation and orientation.
Memory | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  Test of Memory Impairment (T@M). The Test of Memory Impairment (T@M) is a cognitive screening test, with a high discriminatory value for amnestic mild cognitive impairment and mild Alzheimer's disease among the general population. It consists of five sections: Immediate Memory, Temporal Orientation Memory, Semantic Remote Memory, Free Recall Memory and Cue Recall Memory
Functional Status | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  Lawton and Brody Instrumental Activities of Daily Living Scale. It evaluates the daily functionality of the person by means of 8 items: ability to use the telephone, shopping, food preparation, housekeeping, laundry, use of means of transportation and responsibility regarding medication and administration of their finances.
Affectivity and Emotions | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  PANAS questionnaire of positive and negative moods. This questionnaire allows to evaluate, separately, the positive (10 questions) and negative (10 questions) emotional experiences recently lived.
Social network | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  OARS Social Resources Scale. It assesses the social network of the old adults.
Loneliness | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  DeJong Loneliness Questionnaire. Assesses emotional loneliness, missing an intimate relationship, and social loneliness, missing a wider social network.
Acceptance of Technology | Three assessments: (1) Baseline assesment: Month 1, (2) 1st follow-up assessment: between month 7 and month 10; and (3) 2nd follow-up assessment: between month 13 and month 16.
  d-hoc user experience questionnaire based on the Technology Acceptance Model (Nieto-Vietes et al., 2023)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Psychology of the University of Santiago de Compostela, Santiago de Compostela, Galicia
  - Envita Digital Solutions S.L., Vigo, Pontevedra/Galicia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villar F, Serrat R. [Talk to them: Narrative care within a person-centered care framework]. Rev Esp Geriatr Gerontol. 2017 Jul-Aug;52(4):216-222. doi: 10.1016/j.regg.2016.06.004. Epub 2016 Jul 25. Spanish. PMID 27461990
- [Background] Kitwood T, Bredin K. Towards a theory of dementia care: personhood and well-being. Ageing Soc. 1992;12:269-87. doi: 10.1017/s0144686x0000502x. No abstract available. PMID 11654434
- [Background] Costa NP, Polaro SH, Vahl EA, Goncalves LH. Storytelling: a care technology in continuing education for active ageing. Rev Bras Enferm. 2016 Nov-Dec;69(6):1132-1139. doi: 10.1590/0034-7167-2016-0390. English, Portuguese. PMID 27925090
- [Background] Stargatt J, Bhar S, Bhowmik J, Al Mahmud A. Digital Storytelling for Health-Related Outcomes in Older Adults: Systematic Review. J Med Internet Res. 2022 Jan 12;24(1):e28113. doi: 10.2196/28113. PMID 35019845
- [Background] Subramaniam P, Woods B. Digital life storybooks for people with dementia living in care homes: an evaluation. Clin Interv Aging. 2016 Sep 16;11:1263-1276. doi: 10.2147/CIA.S111097. eCollection 2016. PMID 27698556
- [Background] Gately ME, Muccini S, Eggleston BA, McLaren JE. Program Evaluation of My Life, My Story: Virtual Storytelling in the COVID-19 Age. Clin Gerontol. 2022 Jan-Feb;45(1):195-203. doi: 10.1080/07317115.2021.1931610. Epub 2021 Jul 5. PMID 34219605
- [Background] Rios Rincon AM, Miguel Cruz A, Daum C, Neubauer N, Comeau A, Liu L. Digital Storytelling in Older Adults With Typical Aging, and With Mild Cognitive Impairment or Dementia: A Systematic Literature Review. J Appl Gerontol. 2022 Mar;41(3):867-880. doi: 10.1177/07334648211015456. Epub 2021 May 19. PMID 34009053